CLINICAL TRIAL: NCT00774150
Title: Transdisciplinary Studies of CBT for Anxiety in Youth
Brief Title: Transdisciplinary Studies of CBT for Anxiety in Youth: Child Anxiety Treatment Study
Acronym: CATS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Neal Ryan, Joaquim Puig-Antich Professor of Psychiatry, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PRO07110273; P50MH080215-01A1 (NIH)
Record Dates: First submitted 2008-10-16; First posted 2008-10-17 (Estimated); Last update posted 2014-07-18 (Estimated); Status verified 2014-07

CONDITIONS: Generalized Anxiety Disorder; Separation Anxiety Disorder; Social Phobia
Keywords: Neural correlates of pediatric anxiety disorder; Social correlates of pediatric anxiety disorder; Generalized Anxiety Disorder in pediatric populations; Separation Anxiety Disorder in pediatric populations; Social Phobia in pediatric populations
MeSH Terms: conditions — Generalized Anxiety Disorder; Anxiety, Separation; Phobia, Social | interventions — Cognitive Behavioral Therapy; Person-Centered Psychotherapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1. Cognitive Behavioral Therapy (Experimental)
  Interventions: Behavioral: Cognitive Behavioral Therapy
- 2. Client Centered Therapy (Active Comparator)
  Interventions: Behavioral: Client Centered Therapy

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy — 16 sessions of CBT
  Arms: 1. Cognitive Behavioral Therapy
Behavioral: Client Centered Therapy — 16 sessions of CCT
  Arms: 2. Client Centered Therapy

SUMMARY:
The purpose of this study is to investigate neurobehavioral, affective, and social processes that may influence and predict treatment response in pediatric anxiety disorders.

DETAILED DESCRIPTION:
This protocol proposes to study neurobehavioral and social correlates of treatment response in 200 youth (ages 9-13) with general anxiety disorder (GAD), separation anxiety disorder (SAD), and social phobia (SP). All youth with an anxiety disorder will receive 14 weeks of Cognitive Behavioral Therapy (CBT) or Client Centered Therapy (CCT) for child anxiety disorders. The study combines state-of-the-art measures from affective neuroscience, ecologically valid (EMA) measures of mood and behavior in natural environments, and measures of family and social context within a developmentally framed treatment study. The study design focuses on predictors and mechanisms of treatment response. This protocol will test key features of a "vigilance-avoidance" model focusing on hypotheses that pretreatment neural correlates of affective reactivity will predict treatment response and early changes in emotional processing will correlate with clinical response during treatment. In addition, the protocol examines how affective experiences within the family and social context are associated with treatment response and change across treatment, and how these are associated with and interact with neurobehavioral changes in affective functioning. Taken together these aspects of the study will advance understanding of the neurobehavioral, affective, and social processes that underpin treatment response in ways that will inform the design, refinement, and optimal developmental timing of cognitive behavioral treatments, and thus, decrease the morbidity, mortality, and lifetime impairments from these common disorders in youth.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of DSM-IV diagnosis of Generalized Anxiety Disorder (GAD), Separation Anxiety Disorder (SAD), and Social Phobia (SP)

Exclusion Criteria:

* 1. IQ below 70 as assessed by the Wechsler Abbreviated Scale of Intelligence (WASI).

  2. Requires current ongoing treatment with psychoactive medications including anxiolytics and antidepressants.

  3. Acutely suicidal or at risk for harm to self or others. 4. Any motor impairments or eye-hand coordination problems 5. Persons not suited for fMRI procedures including those who have cardiac pacemakers, neural pacemakers, surgical clips in the brain or blood vessels, surgically implanted metal plates, screws or pins, cochlear implants, IUDs, metal braces, or other metal objects in their body, especially in the eye. Dental fillings do not present a problem. Plastic or removable dental appliances do not require exclusion. Pregnancy, determined by pregnancy tests on post-menarcheal females.

  6. History of head injury. 7. Neuromuscular or neurological disorder 8. Vision that is 20/40 and below that cannot be corrected by glasses or contacts.

Specific exclusion criteria for anxious participants includes:

1. Current comorbid diagnosis of: primary major depressive disorder (MDD) (subjects who have primary GAD with co-morbid MDD that is secondary in terms of course and functional impact are not excluded), obsessive-compulsive disorder (OCD), post-traumatic stress disorder (PTSD), conduct disorder, substance abuse or dependence
2. Lifetime diagnosis of autism or Asperger syndrome, bipolar disorder, psychotic depression, schizophrenia, or schizoaffective disorder.

Specific exclusion criteria for controls includes:

1. Any current or lifetime DSM-IV diagnosis.
2. Having a parent with current or lifetime DSM-IV diagnosis of anxiety or mood disorders.

Ages: 9 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 194 (Actual)
Dates: Start 2008-10; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Evidence of therapy effects on anxiety symptoms are established by assessments of clinical status, symptoms, affective style, sleep,parent-child interactions using rating scales, self-report measures, and behavioral observations. | 16 weeks

SECONDARY OUTCOMES:
Cognitive and affective information processing will be measured using fMRI, pupil dilation/eye tracking, and event-related potential (ERP) assessment. | 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Neal D Ryan, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Derived] Westbrook CA, Schlund M, Silk JS, Forbes EE, Ryan ND, Dahl RE, McMakin DL, Kendall PC, Mannarino A, Ladouceur CD. The role of reward-related brain activity in response to treatment and later depression severity: data from a randomized controlled trial in early adolescents with anxiety disorders. Transl Psychiatry. 2025 Aug 16;15(1):286. doi: 10.1038/s41398-025-03388-2. PMID 40818984
- [Derived] Tan PZ, Bylsma LM, Silk JS, Siegle GJ, Forbes EE, McMakin DL, Dahl RE, Ryan ND, Ladouceur CD. Neural indices of performance monitoring are associated with daily emotional functioning in youth with anxiety disorders: An ERP and EMA study. Int J Psychophysiol. 2022 Aug;178:34-42. doi: 10.1016/j.ijpsycho.2022.06.004. Epub 2022 Jun 6. PMID 35679962
- [Derived] Sequeira SL, Silk JS, Ladouceur CD, Hanson JL, Ryan ND, Morgan JK, McMakin DL, Kendall PC, Dahl RE, Forbes EE. Association of Neural Reward Circuitry Function With Response to Psychotherapy in Youths With Anxiety Disorders. Am J Psychiatry. 2021 Apr 1;178(4):343-351. doi: 10.1176/appi.ajp.2020.20010094. Epub 2021 Jan 21. PMID 33472390
- [Derived] Ladouceur CD, Tan PZ, Sharma V, Bylsma LM, Silk JS, Siegle GJ, Forbes EE, McMakin DL, Dahl RE, Kendall PC, Mannarino A, Ryan ND. Error-related brain activity in pediatric anxiety disorders remains elevated following individual therapy: a randomized clinical trial. J Child Psychol Psychiatry. 2018 Nov;59(11):1152-1161. doi: 10.1111/jcpp.12900. Epub 2018 Mar 30. PMID 29603219
- [Derived] Silk JS, Tan PZ, Ladouceur CD, Meller S, Siegle GJ, McMakin DL, Forbes EE, Dahl RE, Kendall PC, Mannarino A, Ryan ND. A Randomized Clinical Trial Comparing Individual Cognitive Behavioral Therapy and Child-Centered Therapy for Child Anxiety Disorders. J Clin Child Adolesc Psychol. 2018 Jul-Aug;47(4):542-554. doi: 10.1080/15374416.2016.1138408. Epub 2016 Mar 16. PMID 26983904